CLINICAL TRIAL: NCT01915160
Title: Technology-Based Tools to Enhance Quality of Care in Mental Health Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R34MH096907-01A1 (NIH)
Record Dates: First submitted 2013-07-01; First posted 2013-08-02 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2012-08

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treatment as usual (Active Comparator): Trauma Focused- Cognitive Behavioral Therapy (TF-CBT)
  Interventions: Behavioral: TF-CBT
- tablet assisted therapy toolkit (Experimental): electronically assisted Trauma Focused-Cognitive Behavioral Therapy (eTF-CBT)
  Interventions: Behavioral: eTF-CBT

INTERVENTIONS:
Behavioral: eTF-CBT — Standard treatment with the edition of in-treatment/session iPad activities.
  Arms: tablet assisted therapy toolkit
Behavioral: TF-CBT — Treatment as usual.
  Arms: treatment as usual

SUMMARY:
Nearly 9 million U.S. children (1 in 8) meet criteria for at least one mental health disorder at any point in time. Effective treatments exist for these disorders, but children and families who seek services rarely receive them; mental health providers need more support in the delivery of these interventions to ensure that children and families are receiving the best quality care. This project aims to improve the delivery of best practices for families who seek mental health care by developing creative, technology-based resources for providers. Once we have completed development of the tablet-based resources, we will conduct a small randomized study with 20 families to examine the feasibility and prepare for a large study to test the effectiveness of the resources.

DETAILED DESCRIPTION:
Efficacious treatments exist for a wide range of psychiatric disorders, but these treatments rarely are delivered with high fidelity in mental health service settings. Research is needed to ensure that these treatments become more accessible in day-to-day clinical care. Innovative, low-cost approaches are essential, particularly in settings where resources are limited. Technological advances have made possible the development of low-cost and highly efficient (i.e., minimal time burden to providers) resources that can be delivered via internet, tablets, Smartphone, and other technologies to improve quality of care. Research is needed to inform these efforts and evaluate the feasibility and utility of this approach. Widespread availability of technology-based resources may represent an important step toward making evidence-based treatment more accessible to children and adults if research supports their utility. Our research team has led the development and evaluation of several e-health and e-learning tools for patients and providers. This has positioned us well to develop and rigorously evaluate a technology-based toolkit to enhance providers' delivery of evidence-based treatment. Trauma-Focused Cognitive Behavioral Therapy (TF-CBT), an empirically supported treatment for children with posttraumatic stress reactions, is widely used by community providers and is ideal for testing the use of technology-based resources because the protocol addresses multiple symptom domains as well as both children and caregivers. We propose to develop and examine the feasibility of a technology-based toolkit for TF-CBT (e-TFCBT) that is designed to enhance the quality, accessibility, and efficacy of treatment. The toolkit will consist of web-based applications that are optimized for use on mobile devices. We conducted an interview of 21 nationally certified trainers in TF-CBT to guide an initial list of resources that are intended to address known problems with fidelity and engagement. Providers will use most of these resources in session to maximize fidelity and enhance child engagement and learning. The resources will be alpha-tested with families and providers and then beta-tested with providers; qualitative data will be used to guide refinements to the toolkit. We will then conduct a feasibility trial with 20 families. Results will provide valuable preliminary data in preparation for a randomized controlled trial to examine the additive benefits of web-accessible resources that assist providers in high-fidelity delivery of evidence-based care.

ELIGIBILITY:
Inclusion Criteria:

* victim of at least one potentially traumatic event (e.g. sexual/physical assault, witnessed violence, disaster, serious accident)
* have at least one symptom on each PTSD symptom cluster (re-experiencing, avoidance, hyperarousal)

Exclusion Criteria:

* exhibits psychotic symptoms (active hallucinations, delusions, impaired thought processes) by caregiver or child
* significant cognitive disabilities, developmental delays, or pervasive developmental disorder
* active suicidal or homicidal ideations
* no consistent caregiver available to participate

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2013-11; Primary Completion 2016-01 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Child Involvement Ratings Scale | post-treatment; will be assessed throughout the course of treatment (expected to be 12-20 weeks in duration for each participant)
  Child engagement will be measured via coding of audiotaped sessions by independent, trained raters who are blind to study purpose and hypotheses. The Child Involvement Ratings Scale (CIRS), a 6-item scale that measures child engagement for each session, will be used. Four "positive" involvement items and two "negative" involvement items are rated for each session on a 6-point scale ("not at all" to "a great deal" present). The positive-involvement items emphasize the extent to which children initiate discussions, demonstrate enthusiasm, self-disclose, and demonstrate understanding. Negative-involvement items address withdrawal or avoidance in treatment. Coders provide ratings based on two 10-min segments of session audiotapes (beginning at min 10 and min 40).
Treatment Adherence Checklist-Revised | post-treatment; will be assessed throughout the course of treatment; an expected duration of 12-20 weeks
  Fidelity to the TF-CBT protocol will be measured via coding of audiotaped treatment sessions by independent, trained raters who are blind to study purpose and hypotheses. Ratings will be completed using the Treatment Adherence Checklist-Revised, a behaviorally specific checklist of TF-CBT provider behavior that we have modified for the current study to ensure relevance to the eTF-CBT condition. This checklist will be used to calculate providers' fidelity to each TF-CBT component. An additional 8 items focus on general therapy skills, not specific to TF-CBT, including establishing an agenda, providing a treatment rationale, and assigning homework. Additional items were created to identify use of eTF-CBT tools to differentiate the two treatment conditions. Two independent raters will listen to tape-recorded treatment session tapes and complete the modified TAC-R to code the presence/absence of specific treatment techniques depicted on the tapes.

SECONDARY OUTCOMES:
Kiddie Schedule for Affective Disorders and Schizophrenia for School Age Children - Present and Lifetime Version (K-SADS-PL PTSD module) | 12-20 weeks
  This is a semi-structured interview that is well-established and widely used. It has been used in numerous TF-CBT RCTs. We also will assess functional impairment in school, social, and family life using the K-SADS-PL instrument.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J Ruggiero, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of SC, Charleston, South Carolina, United States

REFERENCES:
- [Derived] Davidson TM, Bunnell BE, Saunders BE, Hanson RF, Danielson CK, Cook D, Chu BC, Dorsey S, Adams ZW, Andrews AR 3rd, Walker JH, Soltis KE, Cohen JA, Deblinger E, Ruggiero KJ. Pilot Evaluation of a Tablet-Based Application to Improve Quality of Care in Child Mental Health Treatment. Behav Ther. 2019 Mar;50(2):367-379. doi: 10.1016/j.beth.2018.07.005. Epub 2018 Jul 27. PMID 30824252
- [Derived] Ruggiero KJ, Bunnell BE, Andrews Iii AR, Davidson TM, Hanson RF, Danielson CK, Saunders BE, Soltis K, Yarian C, Chu B, Adams ZW. Development and Pilot Evaluation of a Tablet-Based Application to Improve Quality of Care in Child Mental Health Treatment. JMIR Res Protoc. 2015 Dec 30;4(4):e143. doi: 10.2196/resprot.4416. PMID 26717906